CLINICAL TRIAL: NCT03939325
Title: Impact of Different Shock Wave Release Frequencies on Disintegration of Renal Stones in Assuit Urology & Nephrology University Hospital
Brief Title: ESWL on Disintegration of Renal Stones
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed El Taher, M.B.B.CH, Assiut University
Other Study IDs: impact of ESWL in Renal Stones
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- first group: patient who exposed to frequency 60 shock wave per min
  Interventions: Radiation: ESWL
- second group: patient who exposed to frequency 80 shock wave per min
  Interventions: Radiation: ESWL
- third group: patient who exposed to frequency 100 shock wave per min
  Interventions: Radiation: ESWL

INTERVENTIONS:
Radiation: ESWL — The impact of different frequencies on pattern of disintegration of renal stones

SUMMARY:
The impact of different frequencies on pattern of disintegration of renal stones

DETAILED DESCRIPTION:
* Prior to the introduction of extracorporeal shockwave lithotripsy (ESWL) in 1980, the only treatment available for calculi that could not pass through the urinary tract was open surgery. Since then, ESWL has become the preferred tool in the urologist's armamentarium for the treatment of renal stones, , ESWL is minimally invasive, exposes patients to less anaesthesia, and yields equivalent stone-free rates in appropriately selected patients.
* The efficacy of ESWL lies in its ability to pulverize calculi in vivo into smaller fragments, which the body can then expulse spontaneously. Shockwaves are generated and then focused onto a point within the body. The shockwaves propagate through the body with negligible dissipation of energy (and therefore damage) owing to the minimal difference in density of the soft tissues. At the stone-fluid interface, the relatively large difference in density, coupled with the concentration of multiple shockwaves in a small area, produces a large dissipation of energy. Via various mechanisms, this energy is then able to overcome the tensile strength of the calculi, leading to fragmentation. Repetition of this process eventually leads to pulverization of the calculi into small fragments that the body can pass spontaneously and painlessly.
* It is well recognized that the popularity of extracorporeal shock wave lithotripsy (SWL), despite its non-invasive character, has decreased during recent years. This is partly explained by the technological achievements in endoscopy and urologists' enthusiasm for such procedures. Another explanation is that many urologists have been insufficiently successful with SWL. The latter effect might to some extent be a result of the performance of the lithotripter used, but in too many cases, it is evident that the principles of how shock wave lithotripsy should be carried out are poorly appliedical aspect

ELIGIBILITY:
Inclusion Criteria:

* Pelvic and upper ureteric stones
* Stone size less than 2 cm
* Stone density up to 1000 HU

Exclusion Criteria:

* Lower calycle stone
* Stone size 2 cm or more
* Stone denstiy more than 1000
* age group less than 18 y
* uncontrolled hypertension patient and bleeding disorder
* Pregnancy
* Patients with UPJ obstruction, ureteral strictures,
* Congenital anomalies
* Previous stented ureter
* Narrow neck of the calycx less than 30 %

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the outpatient clinic from age 18 years to 70 years old with renal stone who candidate for ESWL
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-05-05 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
stone free rate | 2 weeks
  complete disintegration of renal stones or having clinically insignificant gravel smaller than 2 mm

REFERENCES:
- [Background] Shinde S, Al Balushi Y, Hossny M, Jose S, Al Busaidy S. Factors Affecting the Outcome of Extracorporeal Shockwave Lithotripsy in Urinary Stone Treatment. Oman Med J. 2018 May;33(3):209-217. doi: 10.5001/omj.2018.39. PMID 29896328
- [Background] McClinton S, Cameron S, Starr K, Thomas R, MacLennan G, McDonald A, Lam T, N'Dow J, Kilonzo M, Pickard R, Anson K, Keeley F, Burgess N, Clark CT, MacLennan S, Norrie J; TISU Study Group. TISU: Extracorporeal shockwave lithotripsy, as first treatment option, compared with direct progression to ureteroscopic treatment, for ureteric stones: study protocol for a randomised controlled trial. Trials. 2018 May 22;19(1):286. doi: 10.1186/s13063-018-2652-1. PMID 29788982